CLINICAL TRIAL: NCT02926768
Title: A Phase I/II, Open-Label, Safety, Pharmacokinetic and Efficacy Study of Ascending Doses of Oral CK-101 in Patients With Advanced Solid Tumors
Brief Title: Phase I/II Study of CK-101 in NSCLC Patients and Other Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Checkpoint Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CK-101-101
Record Dates: First submitted 2016-09-29; First posted 2016-10-06 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Diseases; Adenocarcinoma
Keywords: Cancer; Non Small Cell Lung Cancer; EGFR sensitivity mutation; T790M; NSCLC; epidermal growth factor receptor; EGFR; EGFR inhibitor
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Diseases; Adenocarcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daily dose of CK-101 (Experimental): Daily oral dose of CK-101
  Interventions: Drug: CK-101

INTERVENTIONS:
Drug: CK-101 — Phase 1: CK-101 will be administered in escalating dosages in a period of 21-day cycles
  Phase 2: CK-101 will be administered daily

SUMMARY:
CK-101 is a novel, potent, small molecule tyrosine kinase inhibitor (TKI) that selectively targets mutant forms of the epidermal growth factor receptor (EGFR) while sparing wild-type (WT) EGFR. The purpose of the study is to evaluate the pharmacokinetic (PK) and safety profile of oral CK-101; to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of oral CK-101; to assess the safety and efficacy of CK-101 in treatment-naive NSCLC patients known to have activating EGFR mutations and previously treated NSCLC patients known to have the T790M EGFR mutation.

DETAILED DESCRIPTION:
This is a first-in-human, two-part, open-label, safety, pharmacokinetic, and efficacy study of oral CK-101 administered daily in ascending doses in patients with advanced solid tumor cancer, followed by a Phase 2 portion at the recommended Phase 2 dose (RP2D) in previously treated non-small cell lung cancer (NSCLC) patients who have documented evidence of EGFR T790M mutation and have failed treatment with a first-line EGFR inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Measureable disease according to RECIST Version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Minimum age of 18 years
* Adequate hematological, hepatic and renal function
* Written consent on an Institutional Review Board-approved informed consent form prior to any study-specific evaluation
* Histologically or cytologically confirmed diagnosis of one of the following:

  1. Metastatic or unresectable locally advanced NSCLC with documented evidence that the tumor harbors one of the two common EGFR mutations known to be associated with EGFR tyrosine kinase inhibitor (TKI) sensitivity (exon 19 deletion, L858R), either alone or in combination with other EGFR mutations, determined by PCR-based testing of the tumor tissue or plasma sample, and without prior exposure to an EGFR-TKI therapy; OR
  2. Metastatic or unresectable locally advanced NSCLC:

     1. with documented evidence that the tumor harbors an EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q); and
     2. with evidence of radiological disease progression while on a previous continuous treatment with a first-generation EGFR TKI. In addition, other lines of therapy may have been given. All patients must have evidence of radiological disease progression on or following the last treatment administered; and
     3. with documented evidence of EGFR T790M mutation determined by PCR-based testing of the tumor tissue or plasma sample following disease progression on most recent treatment regimen (irrespective of whether this is EGFR TKI or chemotherapy).

Exclusion Criteria:

* Active second malignancy or other prior malignancy treated with chemotherapy less than or equal to 6 months prior to treatment with CK-101
* History of, or evidence of clinically active, interstitial lung disease
* Brain metastases unless asymptomatic, stable and not requiring steroids for at least 2 weeks
* Treatment with prohibited medications
* Any toxicity related to prior treatment must have resolved to Grade 1 or less, with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy
* Certain cardiac abnormalities or history
* Non-study related surgical procedures less than or equal to 14 days prior to CK-101 administration
* Females who are pregnant or breastfeeding.
* Refusal to use adequate contraception for fertile patients (females and males)
* Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical study
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Phase I: Incidence of dose-limiting toxicities (DLTs) | From baseline (first dose) to 28 days after last dose, expected average 6 months
Phase II: Objective response rate (ORR): Defined as the rate of complete responses [CR] or partial responses [PR] per RECIST Version 1.1 as assessed by an independent central review | From baseline (first dose) until disease progression or withdrawal from study, expected average 10 months

SECONDARY OUTCOMES:
Phase II: Evaluation of tumor response based on disease control rate as assessed by RECIST 1.1 | From baseline (first dose) until disease progression or withdrawal from study, expected average 10 months
Phase II: Evaluation of tumor response based on duration of response as assessed by RECIST 1.1 | From baseline (first dose) until disease progression or withdrawal from study, expected average 10 months
Phase II: Evaluation of tumor response based on tumor shrinkage as assessed by RECIST 1.1 | From baseline (first dose) until disease progression or withdrawal from study, expected average 10 months
Phase II: Evaluation of tumor response based on progression free survival as assessed by RECIST 1.1 | From baseline (first dose) until disease progression or withdrawal from study, expected average 10 months
Phase I: Change from baseline in QT/QTc interval | Cycle 1 Day 1 until disease progression or withdrawal from study, expected average 10 months
Phase I: Plasma concentrations of CK-101 following dosing with CK-101 as assessed by area under the curve | Days 1, 8 and 15 of Cycle 1 and Day 1 of Cycle 2
Phase I: Plasma concentrations of CK-101 following dosing with CK-101 as assessed by maximum concentration | Days 1, 8 and 15 of Cycle 1 and Day 1 of Cycle 2
Phase I: Plasma concentrations of CK-101 following dosing with CK-101 as assessed by elimination half-life | Days 1, 8 and 15 of Cycle 1 and Day 1 of Cycle 2

CONTACTS AND LOCATIONS:
Locations (19):
- United States (4):
  - Research Site, Sarasota, Florida
  - Research Site, St Louis, Missouri
  - Research Site, Hackensack, New Jersey
  - Research Site, Nashville, Tennessee
- Research Site, Greenslopes, Queensland, Australia
- New Zealand (3):
  - Research Site, Grafton, Auckland
  - Research Site, Christchurch
  - Research Site, Wellington
- Poland (5):
  - Research Site, Poznan, Greater Poland Voivodeship
  - Research Site, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Research Site, Lublin, Lublin Voivodeship
  - Research Site, Bialystok, Podlaskie Voivodeship
  - Research Site, Szczecin, West Pomeranian Voivodeship
- Thailand (6):
  - Research Site, Pathumwan, Bangkok
  - Research Site, Ratchathewi District, Bangkok
  - Research Site, Bangkok Noi District, Bangkok
  - Research Site, Muang District, Chiang Mai
  - Research Site, Khon Kaen
  - Research Site, Muang, Phitsanulok